CLINICAL TRIAL: NCT00000330
Title: Buprenorphine/Naloxone Treatment for Opioid Dependence-Experiment II-2
Brief Title: Buprenorphine/Naloxone Treatment for Opioid Dependence-Experiment II-2 - 5
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-11160-5; R01DA011160 (NIH); R01-11160-5
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Heroin Dependence; Opioid-Related Disorders
Keywords: Heroin Dependence
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders

INTERVENTIONS:
Drug: Opioid-Related Disorders

SUMMARY:
The purpose of this study is to assess the abuse liability and reinforcing effects of intravenous buprenorphine and buprenorphine/naloxone combinations in heroin-dependent volunteers

DETAILED DESCRIPTION:
not available at this time

ELIGIBILITY:
Inclusion Criteria:

Individuals must be at least 18 yrs of age, currently opioid dependent and must not be seeking treatment. Co-morbid substance abuse or dependence disorders may also be present. Individuals must be healthy despite drug dependency and have a history of IV opioid use.

Exclusion Criteria:

Individuals with evidence of an active Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) Axis I psychiatric disorder (e.g. psychosis, manic-depressive illness, organic psychiatric disorders), significant medical illness (e.g. liver or cardiovascular disease) or pregnant female subjects are excluded from study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1999-10; Primary Completion 1999-11 (Actual); Study Completion 1999-11 (Actual)

PRIMARY OUTCOMES:
Subjective dose estimate
Observed withdrawal rating
Opioid antagonist rating
Pupil diameter
Analog rating scale for drug effects
Drug effect characteristics
Drug/Money Preferences

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Amass, Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Health Sciences Center, Denver, Colorado, United States